CLINICAL TRIAL: NCT05165056
Title: Evaluating the Feasibility and Efficacy of Photobiomodulation Therapy in the Prevention and Management of Radiotherapy-induced Vaginal Toxicity: a Randomized Controlled Trial
Brief Title: Photobiomodulation Therapy in the Prevention and Management of Radiotherapy-induced Vaginal Toxicity
Acronym: GynLight
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other); Hasselt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021/099
Record Dates: First submitted 2021-11-23; First posted 2021-12-21 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Radiotherapy Side Effect; Vaginal Abnormality
Keywords: Photobiomodulation therapy
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Patients allocated to the treatment group will receive institutional standard vaginal care in combined with twice weekly PBMT sessions during the radiotherapy course and until two weeks after the end of radiotherapy.
  Interventions: Device: Intimleds
- Control group (No Intervention): Patients allocated to the control group will receive institutional standard vaginal care.

INTERVENTIONS:
Device: Intimleds — INTIMILEDS® is a photobiomodulation device designed for intravaginal use. It's design permits an irradiation of the whole vaginal wall, the vulva, and the cervix, with a constant intensity.
  Arms: Treatment group

SUMMARY:
This study aims to investigate the effectiveness of photobiomodulation therapy (PBMT) in the prevention and management of radiotherapy-induced vaginal toxicity (RIVT). Therefore, we hypothesize that PBMT can reduce the severity of RIVT in gynecological cancer patients, increasing the patient's QoL and sexual functioning.

DETAILED DESCRIPTION:
The global cancer burden keeps rising, and the accompanied side effects remain a significant concern. This project focuses on one of such complications: radiotherapy-induced vaginal toxicity (RIVT). The use of external and internal radiotherapy in gynecological cancers can severely impact the patient's vaginal function. This influences the patient's quality of life (QoL), as it significantly limits sexual intercourse and further physical examination. Management of RIVT urgently requires a comprehensive approach. Photobiomodulation therapy (PBMT) is a non-invasive form of phototherapy that utilizes visible and/or near-infrared light to trigger a cascade of intracellular reactions. PBMT can be used to improve wound healing, and to reduce pain, inflammation, and edema. Literature shows that PBMT can be used for treating the genitourinary syndrome of menopause as it stimulates the synthesis of collagen and elastin and promotes vasodilation in the vaginal submucosa. To date, no clinical trials have investigated the positive effects of PBMT on RIVT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with endometrial cancer
* Scheduled for external beam radiotherapy (EBRT), intracavitary brachytherapy (BT), or a combination
* Age ≥ 18 years
* Able to comply to the study protocol
* Able to sign written informed consent

Exclusion Criteria:

* Metastatic disease
* Pregnancy
* Diagnosis of vaginal stenosis before radiotherapy (RT)
* Previous pelvic tumor or pelvic RT
* Interruption of RT for more than five sessions
* Severe psychological disorder or dementia.
* Inability to speak and understand Dutch
* Substance abuse patients or patients with medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results as judged by the investigator
* Any condition that is unstable or could affect the safety of the patient and their compliance in the study as judged by the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
CTCAE-score | Baseline
  The physician will score the patient's vaginal dryness, discharge, inflammation, stricture, pain and hemorrhage according to the Common Terminology Criteria for Adverse Events (CTCAE)
CTCAE-score | Two weeks post radiotherapy
  The physician will score the patient's vaginal dryness, discharge, inflammation, stricture, pain and hemorrhage according to the Common Terminology Criteria for Adverse Events (CTCAE)
CTCAE-score | Three months post radiotherapy
  The physician will score the patient's vaginal dryness, discharge, inflammation, stricture, pain and hemorrhage according to the Common Terminology Criteria for Adverse Events (CTCAE)
RIVT symptoms | Baseline
  The patient will score their symptoms (dryness, pruritus, discharge, hemorrhage and a burning sensation) via a numeric rating scale (NRS) ranging from 0 (symptom absent) to 10 (most severe form).
RIVT symptoms | Final radiotherapy session
  The patient will score their symptoms (dryness, pruritus, discharge, hemorrhage and a burning sensation) via a NRS ranging from 0 (symptom absent) to 10 (most severe form).
RIVT symptoms | Two weeks post radiotherapy
  The patient will score their symptoms (dryness, pruritus, discharge, hemorrhage and a burning sensation) via a NRS ranging from 0 (symptom absent) to 10 (most severe form).
RIVT symptoms | Three months post radiotherapy
  The patient will score their symptoms (dryness, pruritus, discharge, hemorrhage and a burning sensation) via a NRS ranging from 0 (symptom absent) to 10 (most severe form).
RIVT symptoms | One year post radiotherapy
  The patient will score their symptoms (dryness, pruritus, discharge, hemorrhage and a burning sensation) via a NRS ranging from 0 (symptom absent) to 10 (most severe form).

SECONDARY OUTCOMES:
Vaginal health index (VHI) | Baseline
  A clinical exam will be performed by the physician to evaluate vaginal elasticity, vaginal secretion, pH, epithelial integrity and moisture. These five parameters will be scored on the on the VHI, from 1 (severe symptoms) to 5 (normal vaginal health). A total score can be calculated by adding the scores of the different parameters
Vaginal health index (VHI) | Two weeks post radiotherapy
  A clinical exam will be performed by the physician to evaluate vaginal elasticity, vaginal secretion, pH, epithelial integrity and moisture. These five parameters will be scored on the on the VHI, from 1 (severe symptoms) to 5 (normal vaginal health). A total score can be calculated by adding the scores of the different parameters
Vaginal health index (VHI) | Three months post radiotherapy
  A clinical exam will be performed by the physician to evaluate vaginal elasticity, vaginal secretion, pH, epithelial integrity and moisture. These five parameters will be scored on the on the VHI, from 1 (severe symptoms) to 5 (normal vaginal health). A total score can be calculated by adding the scores of the different parameters
Pain score | Baseline
  A NRS (0, no pain to 10, the most severe pain) will be used to evaluate the patient's pain level due to the RIVT.
Pain score | Two weeks post radiotherapy
  A NRS (0, no pain to 10, the most severe pain) will be used to evaluate the patient's pain level due to the RIVT.
Pain score | Three months post radiotherapy
  A NRS (0, no pain to 10, the most severe pain) will be used to evaluate the patient's pain level due to the RIVT.
Pain score | One year post radiotherapy
  A NRS (0, no pain to 10, the most severe pain) will be used to evaluate the patient's pain level due to the RIVT.
Quality of Life score | Baseline
  The Female Sexual Function Index (FSFI) is a multidimensional, self-reported questionnaire that evaluates the patient's sexual functioning. The questionnaire consists of 19 questions, divided into six subscales (sexual desire, sexual arousal, lubrication, orgasms, sexual gratification and pain during intercourse). The total score ranges from 2 (severely compromised sexual functioning) to 36 (excellent sexual functioning).
Quality of Life score | Two weeks post radiotherapy
  The European Organization for Research and Treatment for Cancer Quality of Life Questionnaires (EORTC QLQ) will be used to assess the patients' quality of life.
Quality of Life score | Three months post radiotherapy
  The European Organization for Research and Treatment for Cancer Quality of Life Questionnaires (EORTC QLQ) will be used to assess the patients' quality of life.
Quality of Life score | One year post radiotherapy
  The European Organization for Research and Treatment for Cancer Quality of Life Questionnaires (EORTC QLQ) will be used to assess the patients' quality of life.
Sexual functioning score | Baseline
  The Female Sexual Function Index (FSFI) is a multidimensional, self-reported questionnaire that evaluates the patient's sexual functioning. The questionnaire consists of 19 questions, divided into six subscales (sexual desire, sexual arousal, lubrication, orgasms, sexual gratification and pain during intercourse). The total score ranges from 2 (severely compromised sexual functioning) to 36 (excellent sexual functioning).
Sexual functioning score | Two weeks post radiotherapy
  The Female Sexual Function Index (FSFI) is a multidimensional, self-reported questionnaire that evaluates the patient's sexual functioning. The questionnaire consists of 19 questions, divided into six subscales (sexual desire, sexual arousal, lubrication, orgasms, sexual gratification and pain during intercourse). The total score ranges from 2 (severely compromised sexual functioning) to 36 (excellent sexual functioning).
Sexual functioning score | Three months post radiotherapy
  The Female Sexual Function Index (FSFI) is a multidimensional, self-reported questionnaire that evaluates the patient's sexual functioning. The questionnaire consists of 19 questions, divided into six subscales (sexual desire, sexual arousal, lubrication, orgasms, sexual gratification and pain during intercourse). The total score ranges from 2 (severely compromised sexual functioning) to 36 (excellent sexual functioning).
Sexual functioning score | One year post radiotherapy
  The Female Sexual Function Index (FSFI) is a multidimensional, self-reported questionnaire that evaluates the patient's sexual functioning. The questionnaire consists of 19 questions, divided into six subscales (sexual desire, sexual arousal, lubrication, orgasms, sexual gratification and pain during intercourse). The total score ranges from 2 (severely compromised sexual functioning) to 36 (excellent sexual functioning).
Sexual distress score | Baseline
  The multidimensional, self-reported Female Sexual Distress Scale-Revised 2005 (FSDS-R) questionnaire will be used to evaluate the patient's sexual distress. This questionnaire consists of 13 items scored from 0 (never occurring) to 4 (always occurring). A score of 11 or more effectively discriminates between patients with female sexual distress and patients without distress.
Sexual distress score | Two weeks post radiotherapy
  The multidimensional, self-reported Female Sexual Distress Scale-Revised 2005 (FSDS-R) questionnaire will be used to evaluate the patient's sexual distress. This questionnaire consists of 13 items scored from 0 (never occurring) to 4 (always occurring). A score of 11 or more effectively discriminates between patients with female sexual distress and patients without distress.
Sexual distress score | Three months post radiotherapy
  The multidimensional, self-reported Female Sexual Distress Scale-Revised 2005 (FSDS-R) questionnaire will be used to evaluate the patient's sexual distress. This questionnaire consists of 13 items scored from 0 (never occurring) to 4 (always occurring). A score of 11 or more effectively discriminates between patients with female sexual distress and patients without distress.
Sexual distress score | One year post radiotherapy
  The multidimensional, self-reported Female Sexual Distress Scale-Revised 2005 (FSDS-R) questionnaire will be used to evaluate the patient's sexual distress. This questionnaire consists of 13 items scored from 0 (never occurring) to 4 (always occurring). A score of 11 or more effectively discriminates between patients with female sexual distress and patients without distress.
Satisfaction score | Two weeks post radiotherapy
  The patients will be asked to evaluate the general pleasantness and soothing effect of the therapeutic intervention. Furthermore, they will be asked to score their global satisfaction with the therapeutic intervention. The patients will score their satisfaction regarding their treatment on the NRS scale 0 (totally not satisfied) to 10 (very satisfied).
Satisfaction score | Three months post radiotherapy
  The patients will be asked to evaluate the general pleasantness and soothing effect of the therapeutic intervention. Furthermore, they will be asked to score their global satisfaction with the therapeutic intervention. The patients will score their satisfaction regarding their treatment on the NRS scale 0 (totally not satisfied) to 10 (very satisfied).
Satisfaction score | One year post radiotherapy
  The patients will be asked to evaluate the general pleasantness and soothing effect of the therapeutic intervention. Furthermore, they will be asked to score their global satisfaction with the therapeutic intervention. The patients will score their satisfaction regarding their treatment on the NRS scale 0 (totally not satisfied) to 10 (very satisfied).

OTHER OUTCOMES:
General patient-, disease-, and treatment-related information | Baseline
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (e.g. age and smoking history). Information regarding the disease- and treatment-related risk factors will be collected through medical records (e.g., tumour type and stage).
General patient-, disease-, and treatment-related information | Three months post radiotherapy
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (e.g. age and smoking history). Information regarding the disease- and treatment-related risk factors will be collected through medical records (e.g., tumour type and stage).
General patient-, disease-, and treatment-related information | One year post radiotherapy
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (e.g. age and smoking history). Information regarding the disease- and treatment-related risk factors will be collected through medical records (e.g., tumour type and stage).
Cancer relapse or recurrence | One year post radiotherapy
  The posibility of cancer relapse or recurrence will be evaluated using the patients' medical records.
Cancer relapse or recurrence | Two years post radiotherapy
  The posibility of cancer relapse or recurrence will be evaluated using the patients' medical records.
Cancer relapse or recurrence | Three years post radiotherapy
  The posibility of cancer relapse or recurrence will be evaluated using the patients' medical records.
Cancer relapse or recurrence | Four years post radiotherapy
  The posibility of cancer relapse or recurrence will be evaluated using the patients' medical records.
Cancer relapse or recurrence | Five years post radiotherapy
  The posibility of cancer relapse or recurrence will be evaluated using the patients' medical records.
Radiotherapy dose | Final radiotherapy session
  During the delineation for RT planning, a vaginal reference point will be constructed. An anatomical vaginal reference point was defined at the level of the Posterior-Inferior Border of Symphysis (PIBS), plus two points ±2 cm (mid/introitus vagina). For BT extra points were selected for the upper vagina at 12/3/6/9 o'clock, at the vaginal surface and 5 mm depth. Dose reporting to these vaginal reference points will be done and the dose to these reference points will then be correlated with RIVT.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Mebis, Prof. Dr., Principal Investigator — Jessa Hospital
Locations (2):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - Jessa Hospital, Hasselt, Limburg